CLINICAL TRIAL: NCT00275106
Title: Treatment Protocol for T-Cell and B-Precursor Cell Lymphoblastic Lymphoma of the European Inter-group Co-operation on Childhood Non-Hodgkin-Lymphoma (EICNHL)
Brief Title: Prednisolone or Dexamethasone Combined With Chemotherapy in Treating Young Patients With Newly Diagnosed Lymphoblastic Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn due to an excess of toxic deaths
Sponsor: Children's Cancer and Leukaemia Group (Other)
Collaborators: European Inter-group Cooperation on Childhood and Adolescent Non Hodgkin Lymphoma (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CCLG-NHL-2004-08; CDR0000454508 (Registry Identifier: PDQ (Physician Data Query)); EU-20598; CCLG-EURO-LIB-02; EICNHL-ERURO-LB02; EUDRACT-2004-0011861-17
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2008-04

CONDITIONS: Lymphoma
Keywords: stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Leucovorin; Mercaptopurine; Methotrexate; Prednisolone; Thioguanine; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: leucovorin calcium
Drug: mercaptopurine
Drug: methotrexate
Drug: prednisolone
Drug: thioguanine
Drug: vincristine sulfate
Procedure: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as prednisolone and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known whether prednisolone is more effective than dexamethasone when given together with combination chemotherapy in treating lymphoblastic lymphoma.

PURPOSE: This phase III randomized clinical trial is studying prednisolone to see how well it works compared to dexamethasone when given together with combination chemotherapy in treating young patients with newly diagnosed lymphoblastic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the event-free survival of young patients with newly diagnosed lymphoblastic lymphoma treated with induction prednisolone vs dexamethasone.
* Compare the safety of standard maintenance treatment over 18 months vs 24 months in these patients.

Secondary

* Determine prognostic factors highly predicative for treatment failure in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study.

* Cytoreductive prephase: All patients receive methotrexate intrathecally (IT) once on day 1 and prednisolone IV or orally 3 times daily on days 1-7.
* Induction phase (part 1): Patients with T-cell lymphoblastic lymphoma (T-LBL) are randomized to 1 of 2 induction treatment arms. Patients with LBL with an unknown immunophenotype are assigned to arm I. Patients with precursor B-cell lymphoblastic lymphoma (pB-LBL) are assigned to arm II.

  * Arm I (T-LBL or LBL with an unknown immunophenotype): Patients receive prednisolone IV or orally 3 times daily on days 8-28; vincristine IV and daunorubicin hydrochloride IV over 1 hour on days 8, 15, 22, and 29; asparaginase IV over 1 hour on days 12, 15, 18, 21, 24, 27, 30, and 33; and methotrexate IT on days 12 and 33; Patients with CNS involvement receive additional methotrexate IT on days 18 and 27. Patients then proceed to part 2 of the induction phase.
  * Arm II (T-LBL or pB-LBL): Patients receive dexamethasone IV or orally 3 times daily on days 8-28. Patients also receive vincristine, daunorubicin hydrochloride, asparaginase, and methotrexate as in arm I. Patients then proceed to part 2 of the induction phase.
* Induction phase (part 2): Patients receive cyclophosphamide IV over 1 hour on days 36 and 64; cytarabine IV on days 38-41, 45-48, 52-55, and 59-62; oral mercaptopurine on days 36-63; and methotrexate IT on days 45 and 59. Two weeks later, patients proceed to protocol M.
* Protocol M: Patients receive oral mercaptopurine once daily on days 1-56 and high-dose methotrexate IV continuously over 24 hours, and methotrexate IT on days 8, 22, 36, and 50. Patients also receive leucovorin calcium IV 42, 48, and 54 hours after the start of high-dose methotrexate infusion. Patients are then stratified according to stage of disease (I or II vs III or IV). Patients with stage I or II disease proceed directly to maintenance therapy 2 weeks after completion of protocol M. Patients with stage III or IV disease proceed to the re-induction phase 2 weeks after completion of protocol M.
* Re-induction phase: Patients receive dexamethasone IV or orally 3 times daily on days 1-21; vincristine IV and doxorubicin hydrochloride IV over 1 hour on days 8, 15, 22, and 29; asparaginase IV over 1 hour on days 8, 11, 15, and 18; cyclophosphamide IV over 1 hour on day 36; cytarabine IV on days 38-41 and 45-48; oral thioguanine on days 36-49; and methotrexate IT on days 38 and 45. Patients proceed to maintenance therapy 2 weeks after completion of the re-induction phase.
* Maintenance therapy: Patients with T-LBL are randomized to 1 of 2 maintenance treatment arms. Patients with pB-LBL or LBL with an unknown immunophenotype are assigned to arm I. Any patients with evidence of initial CNS involvement undergo cranial radiotherapy before starting maintenance therapy. Patients must show no evidence of progressive disease before starting maintenance therapy.

  * Arm I: Patients receive oral mercaptopurine once a day and oral methotrexate once a week for up to 2 years (from the first day of the cytoreductive phase) in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive treatment as in arm I for up to 1½ years (from the first day of the cytoreductive phase) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: Approximately 600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed lymphoblastic lymphoma (LBL)

  * Stage I-IV disease
  * T-cell LBL, precursor B-cell LBL, or LBL with an unknown immunophenotype

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No known HIV or AIDS infection
* No severe immunodeficiency
* No other prior malignancy
* No prior disease that would preclude treatment with chemotherapy

PRIOR CONCURRENT THERAPY:

* More than 2 months since prior systemic corticosteroids for a duration of > 8 days
* No prior chemotherapy
* No prior radiotherapy
* No prior organ transplant
* No trimethoprim-sulfamethoxazole 6 days before or during methotrexate therapy
* No concurrent participation in another clinical trial

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2004-09; Primary Completion 2009-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Conditional event-free survival

SECONDARY OUTCOMES:
Overall survival
Acute and long-term toxicity
Non-lymphoma-related deaths and early deaths (excluding deaths occurring after second line treatment for failure or relapse)

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Wynn, MD, Study Chair — Royal Manchester Children's Hospital; Tim O.B. Eden, MB, BS, FRCPE, FRCP, FRCPCH, F — The Christie NHS Foundation Trust; Alfred Reiter, MD, Study Chair — University Hospital Erlangen
Locations (22):
- Kinderklinik, Giessen, Germany
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Derived] Landmann E, Burkhardt B, Zimmermann M, Meyer U, Woessmann W, Klapper W, Wrobel G, Rosolen A, Pillon M, Escherich G, Attarbaschi A, Beishuizen A, Mellgren K, Wynn R, Ratei R, Plesa A, Schrappe M, Reiter A, Bergeron C, Patte C, Bertrand Y. Results and conclusions of the European Intergroup EURO-LB02 trial in children and adolescents with lymphoblastic lymphoma. Haematologica. 2017 Dec;102(12):2086-2096. doi: 10.3324/haematol.2015.139162. Epub 2017 Oct 5. PMID 28983060